CLINICAL TRIAL: NCT01047319
Title: A Multinational, Multicenter, Open-label, Single-assignment Extension of the MS-LAQ-302 (BRAVO) Study, to Evaluate the Long-term Safety, Tolerability and Effect on Disease Course of Daily Oral Laquinimod 0.6 mg in Subjects With Relapsing Multiple Sclerosis
Brief Title: A Study to Evaluate the Long-term Safety, Tolerability and Effect of Daily Oral Laquinimod 0.6 mg on Disease Course in Subjects With Relapsing Multiple Sclerosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated RRMS studies as sufficient long term clinical data was collected for the study drug in the relevant dose
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-LAQ-302E; 2009-015815-42 (EudraCT Number)
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis
MeSH Terms: interventions — laquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Laquinimod (Experimental): One capsule containing 0.6 mg laquinimod to be administered orally once daily.
  Interventions: Drug: Laquinimod

INTERVENTIONS:
Drug: Laquinimod — One capsule containing 0.6 mg laquinimod to be administered orally once daily.

SUMMARY:
To make laquinimod 0.6 mg available for all subjects who completed the placebo-controlled MS-LAQ-302 study according to the protocol and to evaluate the long-term safety, tolerability and effect on disease course of daily oral laquinimod 0.6 mg in subjects with relapsing multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have completed the Termination visit of MS-LAQ-302 (completion of all Termination visit activities) according to the MS-LAQ-302 protocol.
2. Women of child-bearing potential must practice an acceptable method of birth control [acceptable methods of birth control in this open label extension phase include: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch (or hormone-releasing vaginal ring), long-acting injectable contraceptive, partner's vasectomy or double-barrier method (condom or diaphragm with spermicide)] during the study and up to 30 days after the last dose of the study drug..
3. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.
4. Subjects must be able to comprehend, sign and date a written informed consent prior to entering the MS-LAQ-302E study.

Exclusion Criteria:

1. Premature discontinuation from the MS-LAQ-302 study, for any reason.
2. Pregnancy [according to urine dipstick β-HCG test performed at Baseline (Month 0E) visit] or breastfeeding.
3. Subjects with clinically significant or unstable medical or surgical condition detected or worsened during the MS-LAQ-302 study, which preclude safe participation and completion of the MS-LAQ-302E study. Acute exacerbation of MS will not exclude participation in the MS-LAQ-302E study.
4. Use of inhibitors of CYP3A4 within 2 weeks prior to baseline visit (V0E, Month 0E).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1047 (Actual)
Dates: Start 2010-05-27 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Timothy Vollmer, MD, Principal Investigator — University of Colorado, Denver
Locations (144):
- United States (22):
  - Teva Investigational Site 1267, Homewood, Alabama
  - Teva Investigational Site 1237, Phoenix, Arizona
  - Teva Investigational Site 1279, Phoenix, Arizona
  - Teva Investigational Site 1276, Tucson, Arizona
  - Teva Investigational Site 1272, Pasadena, California
  - Teva Investigational Site 1238, Sacramento, California
  - Teva Investigational Site 1280, Aurora, Colorado
  - Teva Investigational Site 1282, Sarasota, Florida
  - Teva Investigational Site 1275, Atlanta, Georgia
  - Teva Investigational Site 1250, Peoria, Illinois
  - Teva Investigational Site 1260, Indianapolis, Indiana
  - Teva Investigational Site 1263, Shreveport, Louisiana
  - Teva Investigational Site 1269, Baltimore, Maryland
  - Teva Investigational Site 1273, Albany, New York
  - Teva Investigational Site 1264, Amherst, New York
  - Teva Investigational Site 1261, Akron, Ohio
  - Teva Investigational Site 1245, Cleveland, Ohio
  - Teva Investigational Site 1247, Columbus, Ohio
  - Teva Investigational Site 1244, Portland, Oregon
  - Teva Investigational Site 1281, Nashville, Tennessee
  - Teva Investigational Site 1270, Roanoke, Virginia
  - Teva Investigational Site 1253, Tacoma, Washington
- Bulgaria (17):
  - Teva Investigational Site 5914, Pleven
  - Teva Investigational Site 5915, Pleven
  - Teva Investigational Site 5917, Plovdiv
  - Teva Investigational Site 4212, Rousse
  - Teva Investigational Site 5916, Shumen
  - Teva Investigational Site 5920, Sofia
  - Teva Investigational Site 5907, Sofia
  - Teva Investigational Site 5910, Sofia
  - Teva Investigational Site 5909, Sofia
  - Teva Investigational Site 5919, Sofia
  - Teva Investigational Site 5906, Sofia
  - Teva Investigational Site 5908, Sofia
  - Teva Investigational Site 5911, Sofia
  - Teva Investigational Site 5912, Sofia
  - Teva Investigational Site 5918, Stara Zagora
  - Teva Investigational Site 5913, Varna
  - Teva Investigational Site 4211, Veliko Tarnovo
- Croatia (5):
  - Teva Investigational Site 6003, Osijek
  - Teva Investigational Site 6005, Varaždin
  - Teva Investigational Site 6001, Zagreb
  - Teva Investigational Site 6002, Zagreb
  - Teva Investigational Site 6006, Zagreb
- Czechia (4):
  - Teva Investigational Site 5419, Olomouc
  - Teva Investigational Site 5418, Prague
  - Teva Investigational Site 5420, Praha 5- Motol
  - Teva Investigational Site 5421, Teplice
- Estonia (3):
  - Teva Investigational Site 5508, Kohtla-Järve
  - Teva Investigational Site 5507, Tallinn
  - Teva Investigational Site 5509, Tartu
- Georgia (3):
  - Teva Investigational Site 8102, Tbilisi
  - Teva Investigational Site 8104, Tbilisi
  - Teva Investigational Site 8103, Tbilisi
- Germany (3):
  - Teva Investigational Site 6703, Berlin
  - Teva Investigational Site 6402, Berlin
  - Teva Investigational Site 6400, Ulm
- Israel (2):
  - Teva Investigational Site 8041, Jerusalem
  - Teva Investigational Site 8040, Ramat Gan
- Italy (9):
  - Teva Investigational Site 3056, Bologna
  - Teva Investigational Site 3053, Cefalù
  - Teva Investigational Site 3054, Chieti
  - Teva Investigational Site 3061, Empoli
  - Teva Investigational Site 3049, Florence
  - Teva Investigational Site 3055, Napoli
  - Teva Investigational Site 3048, Rome
  - Teva Investigational Site 3052, Rome
  - Teva Investigational Site 3050, Rome
- Lithuania (2):
  - Teva Investigational Site 5708, Kaunas
  - Teva Investigational Site 5707, Šiauliai
- North Macedonia (3):
  - Teva Investigational Site 6500, Skopje
  - Teva Investigational Site 6501, Skopje
  - Teva Investigational Site 6502, Skopje
- Poland (18):
  - Teva Investigational Site 5337, Bialystok
  - Teva Investigational Site 5329, Gdansk
  - Teva Investigational Site 5338, Gdansk
  - Teva Investigational Site 4213, Gmina Końskie
  - Teva Investigational Site 6602, Gorzów Wielkopolski
  - Teva Investigational Site 5333, Grodzisk Mazowiecki
  - Teva Investigational Site 5334, Katowice
  - Teva Investigational Site 5339, Katowice
  - Teva Investigational Site 6603, Kielce
  - Teva Investigational Site 5332, Kościerzyna
  - Teva Investigational Site 5345, Krakow
  - Teva Investigational Site 5328, Lodz
  - Teva Investigational Site 5330, Olsztyn
  - Teva Investigational Site 5331, Szczecin
  - Teva Investigational Site 5340, Warsaw
  - Teva Investigational Site 5341, Warsaw
  - Teva Investigational Site 5336, Warsaw
  - Teva Investigational Site 5335, Wroclaw
- Romania (9):
  - Teva Investigational Site 5235, Baloteşti
  - Teva Investigational Site 5218, Bucharest
  - Teva Investigational Site 5214, Bucharest
  - Teva Investigational Site 5213, Bucharest
  - Teva Investigational Site 5215, Cluj-Napoca
  - Teva Investigational Site 5217, Constanța
  - Teva Investigational Site 8209, Craiova
  - Teva Investigational Site 5216, Iași
  - Teva Investigational Site 5219, Sibiu
- Russia (11):
  - Teva Investigational Site 5043, Barnaul
  - Teva Investigational Site 5033, Moscow
  - Teva Investigational Site 5041, Moscow
  - Teva Investigational Site 5032, Moscow
  - Teva Investigational Site 5038, Novosibirsk
  - Teva Investigational Site 5042, Novosibirsk
  - Teva Investigational Site 5036, Saint Petersburg
  - Teva Investigational Site 5035, Saint Petersburg
  - Teva Investigational Site 5034, Saint Petersburg
  - Teva Investigational Site 5037, Samara
  - Teva Investigational Site 5044, Ufa
- Slovakia (4):
  - Teva Investigational Site 6200, Bratislava
  - Teva Investigational Site 6201, Bratislava
  - Teva Investigational Site 6202, Nitra
  - Teva Investigational Site 6203, Žilina
- South Africa (7):
  - Teva Investigational Site 9007, Bloemfontein
  - Teva Investigational Site 9001, Cape Town
  - Teva Investigational Site 9004, Johannesburg
  - Teva Investigational Site 9003, Parktown- Johannesburg
  - Teva Investigational Site 9008, Pietermaritzburg
  - Teva Investigational Site 9005, Pretoria
  - Teva Investigational Site 9006, Rosebank
- Spain (7):
  - Teva Investigational Site 3147, Barcelona
  - Teva Investigational Site 3154, Figueres-Girona
  - Teva Investigational Site 3149, L'Hospitalet de Llobregat
  - Teva Investigational Site 3152, Madrid
  - Teva Investigational Site 3151, Málaga
  - Teva Investigational Site 3148, Seville
  - Teva Investigational Site 3153, Tortosa-Tarragona
- Ukraine (15):
  - Teva Investigational Site 6503, Chernihiv
  - Teva Investigational Site 5823, Chernivtsi
  - Teva Investigational Site 5811, Dnipropetrovsk
  - Teva Investigational Site 5812, Donetsk
  - Teva Investigational Site 5814, Ivano-Frankivsk
  - Teva Investigational Site 5817, Kharkiv
  - Teva Investigational Site 5818, Kharkiv
  - Teva Investigational Site 5815, Kharkiv
  - Teva Investigational Site 5822, Kyiv
  - Teva Investigational Site 5809, Lviv
  - Teva Investigational Site 5820, Odesa
  - Teva Investigational Site 5821, Poltava
  - Teva Investigational Site 5810, Vinnytsia
  - Teva Investigational Site 5819, Zaporizhzhya
  - Teva Investigational Site 5816, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who completed the full duration of the double-blind BRAVO study (study MS-LAQ-302) were eligible to enter into Study MS-LAQ-302E. Of the 1090 participants who completed MS-LAQ-302, 1047 opted to continue into the open-label extension study.
Pre-assignment Details: 1047 subjects with RRMS were enrolled to receive laquinimod 0.6 mg daily at 144 study sites in 18 countries by 144 investigators.
Groups:
- Early Laquinimod: All participants in MS-LAQ-302E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Early laquinimod subgroup included participants in MS-LAQ-302 double-blind study who were administered laquinimod 0.6 mg daily for 24 months.
- Switch From Placebo: All participants in MS-LAQ-302E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Switch from placebo subgroup included participants in MS-LAQ-302 double-blind study who were administered placebo daily for 24 months.
- Switch From Avonex: All participants in MS-LAQ-302E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Switch from Avonex subgroup included participants in MS-LAQ-302 rater-blind study who were administered Avonex 30 mcg IM once weekly for 24 months.
Period: Overall Study
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex
Started | 345 | 350 | 352
Completed | 0 | 0 | 0
Not Completed | 345 | 350 | 352
Not completed — Teva requested participant withdrawal | 3 | 0 | 1
Not completed — Protocol Violation | 3 | 2 | 4
Not completed — Lack of Efficacy | 4 | 3 | 3
Not completed — Death | 5 | 1 | 5
Not completed — Pregnancy | 13 | 8 | 8
Not completed — Physician Decision | 12 | 9 | 10
Not completed — Lost to Follow-up | 14 | 10 | 10
Not completed — Adverse Event | 16 | 27 | 21
Not completed — Withdrawal by Subject | 77 | 75 | 87
Not completed — Study terminated by Sponsor | 198 | 215 | 203

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the MS-LAQ-302 extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex | Total
Number analyzed (Participants) | 345 | 350 | 352 | 1047
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.16) | 40.1 (9.23) | 40.1 (9.34) | 39.8 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 245 | 234 | 707
  Male | 117 | 105 | 118 | 340
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Oriental | 1 | 0 | 1 | 2
  Black/African American | 2 | 2 | 2 | 6
  White | 338 | 346 | 348 | 1032
  Unknown | 2 | 2 | 0 | 4
  Other | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event was defined as any untoward medical occurrence that develops or worsens in severity following start of treatment and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs (SAE) include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes. TEAEs associated with cancer, ischemic heart disease, cerebrovascular events, and arthritis were considered to be of special interest.
Time Frame: Day 1 up to 7.13 years
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex
Number analyzed (Participants) | 345 | 350 | 352
Participants
  =>1 TEAE | 290 | 303 | 279
  =>1 Serious TEAE | 54 | 65 | 51
  =>1 Severe TEAE | 36 | 54 | 44
  =>1 TEAE causing discontinuation | 20 | 28 | 23
  =>1 TEAE of special interest | 66 | 64 | 73
  =>1 treatment-related TEAE | 66 | 76 | 96
  =>1 TEAE leading to death | 5 | 3 | 5

2. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Signs
Description: Vital signs with potentially clinically significant abnormal results were evaluated using the following significance criteria:
  * Pulse rate: >=120 and increase >=30 beats/minute
  * Systolic blood pressure low: <=90 and decrease >=30 mmHg
  * Systolic blood pressure high: >=180 and increase >=30 mmHg
  * Diastolic blood pressure low: <=50 and decrease >=20 mmHg
  * Diastolic blood pressure high: >=100 and increase >=20 mmHg
  Note that the change is compared to baseline,
Time Frame: Baseline (Day 0 for extension), Day 1 up to 7.13 years
Population: Safety analysis set of participants with a baseline and post-baseline value for that vital sign,
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex
Number analyzed (Participants) | 345 | 350 | 352
Participants
  Participants with at least one abnormality | 19 | 23 | 19
  Pulse rate - high | 2 | 0 | 0
  Systolic blood pressure - low | 4 | 7 | 9
  Systolic blood pressure - high | 0 | 2 | 0
  Diastolic blood pressure - low | 4 | 5 | 4
  Diastolic blood pressure - high | 9 | 10 | 7

3. Secondary Outcome: Participants With Serum Chemistry Laboratory Tests That Were Potentially Clinically Significant (PCS) Abnormal Comparing Baseline to Any Time During the Study
Description: Counts include two conditions:
  * a change from High / Non-PCS at baseline to Low PCS at any point during the study
  * a change from Low / Non-PCS at baseline to High PCS at any point during the study
  Participants whose condition was not changed from baseline or was changed to a non-PCS value are included in the population count.
  ALT=alanine aminotransferase ALP=alkaline phosphatase P-amylase=amylase, pancreatic AST=aspartate aminotransferase CRP=C reactive protein CK=creatine kinase CTN=creatinine FIB=fibrinogen GGT=gamma glutamyl transferase K=potassium
Time Frame: Baseline (Day 0), Day 1 to 7.13 years
Population: Safety analysis set of participants with both a baseline and a post-baseline value for the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex
Number analyzed (Participants) | 344 | 349 | 347
Participants
  ALT - change from Low / Non-PCS to High PCS | 5 | 8 | 10
  Albumen - change from High / Non-PCS to Low PCS | 0 | 1 | 0
  ALP - change from Low / Non-PCS to High PCS | 0 | 2 | 0
  p-Amylase - change from Low / Non-PCS to High PCS | 5 | 1 | 2
  AST - change from Low / Non-PCS to High PCS | 3 | 2 | 5
  Bilirubin - change from Low / Non-PCS to High PCS | 2 | 3 | 2
  CRP - change from Low / Non-PCS to High PCS | 36 | 32 | 31
  Calcium - change from High / Non-PCS to Low PCS | 1 | 1 | 1
  Calcium - change from Low / Non-PCS to High PCS | 1 | 1 | 2
  CK - change from Low / Non-PCS to High PCS | 11 | 12 | 10
  CTN - change from Low / Non-PCS to High PCS | 1 | 1 | 0
  FIB - change from Low / Non-PCS to High PCS | 22 | 24 | 25
  GGT - change from Low / Non-PCS to High PCS | 16 | 22 | 18
  Glucose - change from High / Non-PCS to Low PCS | 12 | 16 | 11
  Glucose - change from Low / Non-PCS to High PCS | 4 | 5 | 2
  Phosphate-change from High / Non-PCS to Low PCS | 12 | 12 | 6
  Phosphate-change from Low / Non-PCS to High PCS | 17 | 18 | 16
  K - change from High / Non-PCS to Low PCS | 2 | 4 | 2
  K - change from Low / Non-PCS to High PCS | 46 | 39 | 38
  Sodium - change from High / Non-PCS to Low PCS | 4 | 2 | 3
  Sodium - change from Low / Non-PCS to High PCS | 21 | 16 | 17
  Urea - change from Low / Non-PCS to High PCS | 4 | 4 | 3

4. Secondary Outcome: Participants With Serum Hematology Laboratory Tests That Were Potentially Clinically Significant (PCS) Abnormal Comparing Baseline to Any Time During the Study
Description: Counts include two conditions:
  * a change from High / Non-PCS at baseline to Low PCS at any point during the study
  * a change from Low / Non-PCS at baseline to High PCS at any point during the study
  Participants whose condition was not changed from baseline or was changed to a non-PCS value are included in the population count.
Time Frame: Baseline (Day 0), Day 1 to 7.13 years
Population: Safety analysis set of participants with both a baseline and a post-baseline value for the test.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex
Number analyzed (Participants) | 344 | 349 | 347
Participants
  Hematocrit - change from High / Non-PCS to Low PCS | 30 | 25 | 21
  Hemoglobin -change from High / Non-PCS to Low PCS | 21 | 24 | 15
  Leukocytes - change from High / Non-PCS to Low PCS | 2 | 4 | 2
  Leukocytes - change from Low / Non-PCS to High PCS | 4 | 1 | 5
  Neutrophils - change from High/Non-PCS to Low PCS | 25 | 12 | 14
  Platelets - change from High / Non-PCS to Low PCS | 5 | 3 | 2
  Platelets - change from Low / Non-PCS to High PCS | 4 | 4 | 4

5. Secondary Outcome: Participants With Electrocardiogram (ECG) Fiindings That Shifted From Baseline to Any Time During the Study
Description: Shifts are presented as Baseline finding / Worse finding at anytime during the study.
  Categories for findings are:
  * normal
  * abnormal, not clinically significant (Not CS)
  * abnormal, clinically significant (CS)
Time Frame: Baseline (Day 0), Day 1 to 7.13 years
Population: Safety analysis set of participants with both a baseline and a post-baseline ECG.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex
Number analyzed (Participants) | 340 | 346 | 345
Participants
  Normal / Normal | 150 | 148 | 134
  Normal / Abnormal, Not CS | 109 | 125 | 119
  Normal / Abnormal, CS | 5 | 3 | 5
  Abnormal, Not CS / Normal | 5 | 7 | 20
  Abnormal, Not CS / Abnormal, Not CS | 67 | 62 | 64
  Abnormal, Not CS / Abnormal, CS | 4 | 0 | 2
  Abnormal, CS / Normal | 0 | 0 | 0
  Abnormal, CS / Abnormal, Not CS | 0 | 0 | 1
  Abnormal, CS / Abnormal, CS | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 7.13 years
Groups:
- Early Laquinimod: All participants in MS-LAQ- 302E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Early laquinimod subgroup included participants in MS-LAQ-302 double-blind study who were administered laquinimod 0.6 mg daily for 24 months.
- Switch From Placebo: All participants in MS-LAQ- 302E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped.
  The Switch from Placebo subgroup included participants in MS-LAQ-302 double-blind study who were administered placebo daily for 24 months.
- Switch From Avonex: All participants in MS-LAQ- 302E were administered 1 capsule containing laquinimod 0.6 mg taken orally at the same hour every day until the product was commercially available or development stopped. The Switch from Avonex subgroup included participants in MS-LAQ-302 rater-blind study who were administered Avonex 30 mcg IM once weekly for 24 months.
Arm/Group | Early Laquinimod | Switch From Placebo | Switch From Avonex
All-Cause Mortality (participants affected / at risk) | 5/345 | 3/350 | 5/352
Serious Adverse Events (participants affected / at risk) | 54/345 | 65/350 | 51/352
Other Adverse Events (participants affected / at risk) | 215/345 | 205/350 | 194/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Laquinimod (N=345) | Switch From Placebo (N=350) | Switch From Avonex (N=352)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy to metals (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Incision site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (4) | 3 (3)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Crush syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (4) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cervix disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 4 (5) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bartholin's cyst removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Fracture reduction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Osteosynthesis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Radical hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Splenectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Laquinimod (N=345) | Switch From Placebo (N=350) | Switch From Avonex (N=352)
Anaemia (Blood and lymphatic system disorders) | 22 (34) | 20 (24) | 15 (18)
Bronchitis (Infections and infestations) | 24 (26) | 23 (29) | 16 (27)
Influenza (Infections and infestations) | 27 (34) | 25 (38) | 22 (32)
Nasopharyngitis (Infections and infestations) | 52 (96) | 46 (77) | 37 (58)
Pharyngitis (Infections and infestations) | 11 (18) | 18 (24) | 11 (15)
Respiratory tract infection viral (Infections and infestations) | 20 (25) | 15 (24) | 16 (20)
Upper respiratory tract infection (Infections and infestations) | 36 (62) | 36 (63) | 28 (59)
Urinary tract infection (Infections and infestations) | 22 (30) | 18 (22) | 17 (22)
C-reactive protein increased (Investigations) | 19 (25) | 17 (23) | 14 (16)
Weight increased (Investigations) | 19 (23) | 11 (11) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (27) | 23 (27) | 28 (38)
Back pain (Musculoskeletal and connective tissue disorders) | 49 (74) | 49 (72) | 50 (73)
Headache (Nervous system disorders) | 44 (84) | 60 (121) | 74 (128)
Depression (Psychiatric disorders) | 26 (26) | 20 (21) | 17 (21)
Hypertension (Vascular disorders) | 18 (22) | 21 (23) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT01047319/Prot_SAP_000.pdf